CLINICAL TRIAL: NCT00285155
Title: Assessment of Bupropion on Cognitive Function and Behaviour in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UF7759
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2007-08-09 (Estimated); Status verified 2007-08

CONDITIONS: Healthy
Keywords: bupropion; repeated dose; healthy volunteers; cognitive function; behaviour; tolerance; Persons
MeSH Terms: conditions — Behavior | interventions — Bupropion

INTERVENTIONS:
Drug: Bupropion

SUMMARY:
To evaluate the effects of a 14-day repeated dose of 150 mg bupropion (therapeutic dose) on cognitive and executive functions, behaviour and subjective feelings, after sleep deprivation in 12 healthy male subjects.

DETAILED DESCRIPTION:
The aim of this controlled double-blind randomized 3-session cross-over designed study is to evaluate the effects of a single dose of 150 mg and a 14-day repeated dose of 300 mg bupropion (therapeutic dose) on cognitive and executive functions, behaviour and subjective feelings, and some physical parameters after sleep deprivation in 12 trained healthy volunteers (18-35 years old).

Cognitive and executive functions were assessed by reaction times, critical flicker fusion test, Stroop test, digit symbol substitution test, span test and short term recal of pictures, tapping and tracking tests.

Behaviour and subjective effects explored were :

* feelings frequently experienced with psychotropic drugs assessed by ARCI,
* some mood states as tension, depression, anger, vigor, fatigue and confusion assessed by both POMS and Norris visual analogic scales,
* sleep assessed by LSEQ,
* feeding behaviour assessed by food intake during a meal test and self-ratings of appetite and satiety,

Physical parameters were :

* rest and orthostatic blood pressure and heart rate,
* body temperature and weight.

Bupropion was tested versus both placebo and 20 mg methylphenidate as positive control. Each subject received the 3 treatments, sequently randomized, with a 17-day wash-out period between sessions. Each session was organized as follow :

* 2 20-hour hospitalisations consisting in adverse effects review, physical examination, test training, sleep deprivation, drug compliance evaluation, drug dosing and dispensation, and assessments described above,
* 2 visits consisting in adverse effects review, drug compliance evaluation and drug dispensation.

The total duration of participation for the subjects was 106 days.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 20.0 and 25.00
* no smoker

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2004-11; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Cognitive and executive functions after the first dose and the 14-day treatment.Subjective feelings after the first dose and the 14-day treatment : ARCI, Norris and POMS scales.

SECONDARY OUTCOMES:
Sleep questionnaire after the 14-day treatment. Energy intake after the 14-day treatment. Blood pressure after one dose and the 14-day treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre PETIT, MD-PhD, Principal Investigator — Centre d'Investigation Clinique
Locations (1):
- Centre d'Investigation Clinique, Montpellier, France

REFERENCES:
- [Derived] Chevassus H, Farret A, Gagnol JP, Poncon CA, Costa F, Roux C, Galtier F, Petit P. Psychological and physiological effects of bupropion compared to methylphenidate after prolonged administration in healthy volunteers (NCT00285155). Eur J Clin Pharmacol. 2013 Apr;69(4):779-87. doi: 10.1007/s00228-012-1418-z. Epub 2012 Oct 9. PMID 23052417